CLINICAL TRIAL: NCT05761691
Title: Does Treating Early Childhood Caries Under Local or General Anesthesia Have Varying Effects on OHRQoL: A Randomized Controlled Trial
Brief Title: Does Treating Early Childhood Caries Under Local or General Anesthesia Have Varying Effects on OHRQoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Mohammad Abdullah Alwadaani, Pediatric Dental Resident, Riyadh Elm University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FBGRP-2021-562-421-415
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Oral Health Related Quality of Life OHRQoL
Keywords: Early Childhood Caries; Children; Oral Health-Related Quality of Life; OHRQoL; Dental General Anesthesia; Local Anesthesia
MeSH Terms: interventions — Dental Care

STUDY DESIGN:
Intervention Model Description: Two armed RCT was planned.
  First: children received dental treatment under general anesthesia (Study group)
  Second: Children received dental treatment under local anesthesia (Control group) in regular dental sitting.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children treated for Early childhood caries under general anesthesia (DGA) (Experimental): GA group (Study group) the dental treatment was provided as a day care surgery under general anasthesia for healthy child patients.
  Interventions: Procedure: Dental treatment
- Children treated for Early childhood caries under Local anesthesia (LA) (Experimental): LA goup (control group) the average number of dental visits was required to finish the treatment plan in local anasthesia group around five to six visits.
  Interventions: Procedure: Dental treatment

INTERVENTIONS:
Procedure: Dental treatment — Children treated for ECC under general (DGA) and local anesthesia (LA).

SUMMARY:
A two-arm randomized control trial is to compare the changes in OHRQoL scores among children treated for ECC under general (DGA) and local anesthesia (LA). Outcome variable was OHRQoL, measured using the early childhood oral health impact scale ECOHIS and explanatory variable was the administration of local or general anesthesia.

DETAILED DESCRIPTION:
Ethical Approval:

The study proposal was registered with the research center at Riyadh Elm University (REU), Riyadh, Saudi Arabia, and ethical approval was obtained from the institutional review board (IRB). Informed consent was obtained from the parents of all participants and the data was managed such that complete confidentiality of the patient was maintained. The current study abides by the regulations presented at the Helsinki declaration.

Sample size calculation:

The sample size required to reject the null hypothesis was estimated using the data from a previous study42 wherein 33.3% of the children with treatment under DGA were reported with better OHRQoL in contrast to 3.3% in the control group. With the alpha set at 0.05, the 80% power of study, and the addition of 30% dropout rate, a sample size of a minimum of 50 children in each group was estimated.

Sample selection criteria:

Arab children aged six years or younger, who were recommended for comprehensive dental treatment at Riyadh Elm university hospitals (Munseah and Numthjiah campuses) by pediatric dentistry residents, and who consented to be part of the study were recruited. Before subjecting the recruited participants to randomization, the intraoral findings were documented, radiographs were taken, and a plan of treatment was designed. Children with systemic disease, physical and mental disability, and congenital defect such as amelogenesis imperfecta or cleft lift/palate were excluded.

Study variables:

The OHRQoL was measured using the Arabic version of the Early childhood impact scale ECOHIS.35 This scale has 13 questions and is divided into the child and family impacts. The child impact part includes nine questions under four fields: child OH symptoms, function, psychology and self-image, and social interaction while the family impact part contains four questions under two domains: parental distress and family function.35 Parents responded to the questions on a 6-point Likert scale (0, never; 1, hardly ever; 2, occasionally; 3, often; 4, very often; and 5, do not know). The overall score was calculated by summing the scores of each item and domain separately. Lower scores indicated better OHRQoL

Explanatory variables:

The primary explanatory variable was the administration of local or general anesthesia to perform the comprehensive dental treatment which included pulp therapy, restoration, and extraction of primary teeth. Age and gender of children, family socio-economic status, parent's education level, dental index "dft" decayed and filled teeth, along with fractured and traumatized teeth were also recorded. The details related to clinical examination, dental history, and treatment provided were recorded from the electronic file system "DENTPLUS" at REU hospitals. The average number of dental visits was required to finish the treatment plan in LA group around five to six while in GA group the treatment was provided as a day care surgery for healthy child patients.

Data collection process:

The data collection was carried out from April 2021 to January 2022. During the Child's first appointment, an oral examination was conducted, followed by a comprehensive treatment plan. Additionally, the child's behavior was assessed using the Frankel behavior rating scale before subjecting them to randomization.Each eligible child with no behavioral issues was subjected to a flip coin randomization process and assigned accordingly into the LA or DGA group. The process of flip coin method to assign the children into two groups was carried out until one group reached the required sample size of 50, and then the remaining eligible children were assigned to the subsequent group. Importantly, therapy under LA was planned for children whose parents were fearful and did not consent for DGA. Also, therapy under DGA was planned for children whose parents wanted to complete the treatment in a single session. These children who could not be subjected to randomization process were treated but not included in the study.

In this study, due to obvious reasons, the child-parent duo and the primary investigator performing the dental treatment could not be blinded to the intervention. However, to somewhat follow the blinding process, the primary investigator asked a trained dental auxiliary staff, who was not part of the study, to administer the ECOHIS questionnaire and collect the socio-demographic data. This process where the primary investigator was blinded to the assessment of the outcome variable was followed at the baseline, one week, and one-month data collection timelines. The person carrying out the statistical analyses was blinded to the intervention and the outcome assessment. All the data was first entered in the Microsoft Excel and then transferred to SPSS version 24 (IBM, USA) for data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Arab children
* Age six years or younger

Exclusion Criteria:

* Children systemic disease
* Children with physical and mental disability
* Children with congenital dental defect such as amelogenesis imperfecta
* Children with cleft lift/palate

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male & Female
Enrollment: 73 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Oral health related quality of life OHRQoL | One year
  Oral health related quality of life OHRQoL was measured using the Arabic version of the Early childhood impact scale ECOHIS. This scale has 13 questions and is divided into the child and family impacts. The child impact part includes nine questions under four fields: child OH symptoms, function, psychology and self-image, and social interaction while the family impact part contains four questions under two domains: parental distress and family function. Parents responded to the questions on a 6-point Likert scale (0, never; 1, hardly ever; 2, occasionally; 3, often; 4, very often; and 5, do not know). The overall score was calculated by summing the scores of each item and domain separately with maximum value at (65) . Lower scores indicated better OHRQoL

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Alwadaani, MSc, Principal Investigator — Riyadh Elm University
Locations (1):
- Riyadh Elm University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alwadani MA, Alsulaiman DA, Kakti A, Alamoudi S, Tadakamadla SK, Quadri MFA. Comparison of Oral Health-Related Quality of Life scores in children treated for early childhood caries under general and local anesthesia: a quasi-experimental study. Eur Arch Paediatr Dent. 2023 Dec;24(6):719-728. doi: 10.1007/s40368-023-00835-w. Epub 2023 Aug 29. PMID 37644356

DOCUMENTS (2):
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05761691/SAP_000.pdf
  • Informed Consent Form (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05761691/ICF_001.pdf